CLINICAL TRIAL: NCT04129502
Title: A Randomized Phase 3 Multicenter Open-Label Study to Compare the Efficacy of TAK-788 as First-Line Treatment Versus Platinum-Based Chemotherapy in Patients With Non-Small Cell Lung Cancer With EGFR Exon 20 Insertion Mutations
Brief Title: TAK-788 as First-Line Treatment Versus Platinum-Based Chemotherapy for Non-Small Cell Lung Cancer (NSCLC) With EGFR Exon 20 Insertion Mutations
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-788-3001; NL20191212 (Registry Identifier: CCMO); 2019-001845-42 (Registry Identifier: EudraCT); U1111-1232-6059 (Other Grant/Funding Number: WHO); jRCT2071210098 (Registry Identifier: jRCT)
Record Dates: First submitted 2019-10-07; First posted 2019-10-16 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mobocertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-788 Group (Arm A) (Experimental): TAK-788 160 milligram (mg) with or without food, capsules, orally, once daily until the participants experience PD as assessed by blinded IRC, intolerable toxicity, or another discontinuation criteria.
  Interventions: Drug: TAK-788
- Platinum-based Chemotherapy Group (Arm B) (Active Comparator): Pemetrexed 500 milligram per meter square (mg/m^2) plus cisplatin 75 mg/m^2, infusion, IV, once on Day 1 of 21-day cycle pemetrexed 500 mg/m^2 plus carboplatin, infusion, IV, once at a dose calculated to produce area under curve (AUC) of 5 milligram*minute per milliliter (mg*min/mL) on Day 1 of 21-day cycle until the participants experience PD as assessed by blinded IRC, intolerable toxicity, or another discontinuation criteria. Pemetrexed/cisplatin or pemetrexed/carboplatin will be repeated every 3 weeks for 4 cycles, followed by maintenance treatment with pemetrexed 500 mg/m^2, on Day 1 of a 21-day cycle thereafter.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: TAK-788 — TAK-788 capsule
  Other Names: AP32788; Mobocertinib
  Arms: TAK-788 Group (Arm A)
Drug: Pemetrexed — Pemetrexed IV infusion
  Other Names: Alimta
  Arms: Platinum-based Chemotherapy Group (Arm B)
Drug: Cisplatin — Cisplatin IV infusion
  Arms: Platinum-based Chemotherapy Group (Arm B)
Drug: Carboplatin — Carboplatin IV infusion
  Arms: Platinum-based Chemotherapy Group (Arm B)

SUMMARY:
The purpose of this study is to compare effectiveness of TAK-788 as first-line treatment with that of platinum-based chemotherapy in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) whose tumors has epidermal growth factor receptor (EGFR) exon 20 insertion mutations.

Participants will be randomly assigned to one of the two treatment groups- TAK-788 group or Platinum-based chemotherapy group.

Participants will receive TAK-788 orally and pemetrexed/cisplatin or pemetrexed/carboplatin via vein until the participants experience worsening disease (PD) as assessed by blinded independent review committee (IRC), intolerable harmful effects or another discontinuation criteria.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-788. TAK-788 is being tested to evaluate the efficacy as a first line treatment compare with platinum-based chemotherapy in the participants with locally advanced or NSCLC whose tumors harbor EGFR exon 20 insertion mutations.

The study will enroll approximately 318 patients. Participants will be randomly assigned to one of the two treatment groups-

* TAK-788 Group (Arm A)
* Platinum-based Chemotherapy Group (Arm B)

The participants will be administered with TAK-788 orally in arm A and pemetrexed/cisplatin or pemetrexed/carboplatin intravenously (IV) in arm B until the participants experience progressive disease (PD) as assessed by blinded independent review committee (IRC), intolerable toxicity or another discontinuation criteria. Participants in the chemotherapy group may cross over to treatment with TAK-788 after IRC-assessed PD is documented. Randomized treatment with TAK-788 or platinum-based chemotherapy may be continued after PD, at the discretion of the investigator and with the sponsor's approval, if there is still evidence of clinical benefit.

This multi-center trial will be conducted in United States (US), Europe, and Asia. The overall time to participate in this study is until 3 years after the last participant is randomized. Participants will make multiple visits to the clinic and will be followed for survival, subsequent anticancer therapy, subsequent disease assessment outcome until disease progression on a subsequent anticancer therapy, and participant-reported health status (EuroQoL-5 Dimensions-5 Levels [EQ-5D-5L]) for 3 years after the last participant is randomized in the study and 30 days after the last dose of study drug for safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients (aged 18 years or older)
* Histologically or cytologically confirmed nonsquamous cell locally advanced not suitable for definitive therapy, recurrent, or metastatic (Stage IV) NSCLC
* Documented epidermal growth factor receptor (EGFR) in-frame exon 20 insertion mutation assessed by a clinical laboratory improvements amendment (CLIA)-certified (US sites) or an accredited (outside of the US) local laboratory The EGFR exon 20 insertion mutation can be either alone or in combination with other EGFR or human epidermal growth factor receptor 2 (HER2) mutations except EGFR mutations for which there are approved anti-EGFR tyrosine kinase inhibitors [TKIs] (ie, exon 19 del, L858R, T790M, L861Q, G719X, or S768I, where X is any other amino acid)
* Adequate tumor tissue available, either from primary or metastatic sites, for central laboratory confirmation of EGFR exon 20 insertion mutation
* At least 1 measurable lesion per RECIST Version 1.1
* Life expectancy ≥3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate organ and hematologic function as defined by blood transfusions with a recommended >/ 14 day washout period.

Exclusion Criteria:

* Received prior systemic treatment for locally advanced or metastatic disease, including local administration, such as intra-pleural injection of anticancer medication with the exception noted below:

  * Neoadjuvant or adjuvant chemotherapy/immune therapy for Stage I to III or combined modality chemotherapy/radiation for locally advanced disease is allowed if completed >6 months before the development of metastatic disease.
* Received radiotherapy ≤14 days before randomization or has not recovered from radiotherapy-related toxicities
* Received a moderate or strong cytochrome P450 (CYP)3A inhibitor or moderate or strong CYP3A inducer within 10 days before first dose of TAK-788
* Have been diagnosed with another primary malignancy other than NSCLC
* Have current spinal cord compression or leptomeningeal disease
* Have uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure
* Received a live vaccine within 4 weeks before randomization per Summary of product characteristics (SmPCs) for pemetrexed, cisplatin, and carboplatin
* Taking medication(s) known to be associated with the development of torsades de pointes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Blinded Independent Review Committee (IRC) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to approximately 40 months after the first participant is randomized
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for progressive disease (PD) according to RECIST Version 1.1 are met or death, whichever occurs first.

SECONDARY OUTCOMES:
Confirmed Objective Response Rate (ORR) as Assessed by Blinded Independent Review Committee (IRC) per RECIST Version 1.1 | Up to approximately 40 months after the first participant is randomized
  Confirmed ORR is defined as the percentage of participants who are confirmed to have achieved complete response (CR) or partial response (PR). Confirmed responses are responses that persist on repeat imaging ≥4 weeks after initial response.
Overall Survival (OS) | Up to approximately 40 months after the first participant is randomized
  OS is defined as the interval from the date of randomization until death.
Progression Free Survival (PFS) as Assessed by the Investigator | Up to approximately 40 months after the first participant is randomized
  PFS is defined as the time interval from the date of randomization until the first date at which the criteria for PD according to RECIST Version 1.1 are met or death, whichever occurs first.
Confirmed Objective Response Rate (ORR) as Assessed by the Investigator | Up to approximately 40 months after the first participant is randomized
  Confirmed ORR is defined as the percentage of participants who are confirmed to have achieved CR or PR. Confirmed responses are responses that persist on repeat imaging ≥4 weeks after initial response.
Duration of Response, as Assessed by the Blinded Independent Review Committee (IRC) and the Investigator | Up to approximately 40 months after the first participant is randomized
  Duration of response is defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that PD or death (whichever occurs first) is objectively documented.
Time to Response, as Assessed by the Blinded Independent Review Committee (IRC) and the Investigator | Up to approximately 40 months after the first participant is randomized
  Time to response is defined as the time interval from the date of randomization until the initial observation of CR or PR.
Disease Control Rate (DCR) as Assessed by the Blinded Independent Review Committee (IRC) and the Investigator | Up to approximately 40 months after the first participant is randomized
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) (in the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks) after the initiation of study drug.
Patient-reported Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 | Up to approximately 40 months after the first participant is randomized
  EORTC QLQ-C30 is a cancer-specific questionnaire which comprises of 5 functional scales (physical, role, cognitive, emotional, and social functioning); 3 symptom scales (fatigue, pain, and nausea/vomiting); and a global health status/quality-of-life (QoL) scale. Six single-item scales are also included (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Raw scores will be converted into scale scores ranging from 0 to 100. For the functional scales and the global health status/QoL scale, higher scores represent better HRQoL, whereas for the symptom scales lower scores represent better HRQoL (i.e., a low level of symptomatology/problems).
Participant-reported Symptoms as Assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire, Lung Cancer Module (QLQ-LC13) | Up to approximately 40 months after the first participant is randomized
  EORTC QLQ-LC13 is a cancer-specific questionnaire which comprises of 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and use of pain medication. Raw scores will be converted into scale scores ranging from 0 to 100. Higher scores represent a high level of symptomatology/problems.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (134):
- United States (11):
  - City of Hope National Medical Center, Long Beach, California
  - University of California Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - AdventHealth, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center - 330 Brookline Ave, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
- Australia (3):
  - GenesisCare North Shore, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
- Klinik Floridsdorf, Vienna, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - Grand Hopital de Charleroi asbl, Charleroi, Hainaut
  - AZ Sint-Lucas, Aalst, Oost-Vlaanderen
- Canada (4):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Du Sacre Coeur de Montreal, Montreal, Quebec
- China (12):
  - Beijing Cancer Hospital - PPDS, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Beijing Cancer Hospital - PPDS, Beijing
  - Beijing Chest Hospital, Capital Medical Univerity, Beijing
  - Icahn School of Medicine at Mount Sinai, Beijing
  - Sichuan Cancer Hospital & Institute, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Tumor Hospital, Harbin
  - Shanghai East Hospital, Shanghai
  - Hubei Cancer Hospital, Wuhan
- France (11):
  - Centre Francois Baclesse, Caen, Calvados
  - CHU de Nantes - Hoptal Nord Laennec, Nantes, Loire-Atlantique
  - Hopital Calmette, Lille, Nord
  - Centre Leon Berard, Lyon, Rhone
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - CHU de Grenoble, Grenoble
  - Hopital Nord AP-HM, Marseille
  - CRLC Val d'Aurelle - Paul Lamarque, Montpellier
  - Hopital Tenon, Paris
  - Nouvel Hopital Civil, Strasbourg
  - Hopital Larrey, Toulouse
- Germany (6):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - LMU Klinikum der Universitat Munchen, München, Bavaria
  - University Clinic Regensburg, Regensburg, Bavaria
  - Universitatsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Helios Klinikum Emil Von Behring, Berlin
- Greece (2):
  - Sotiria Chest Hospital of Athens, Athens, Attica
  - Bioclinic Thessaloniki (Galinos clinic), Thessaloniki
- Hong Kong (6):
  - Princess Margaret Hospital, Kowloon City, Kowloon City
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Elizabeth Hospital (QEH), Hong Kong
  - Queen Mary Hospital - PPDS, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Israel (2):
  - Soroka University Medical Centre, Beersheba
  - Sheba Medical Center - PPDS, Ramat Gan
- Italy (9):
  - AORN Dei Colli- Ospedale Monaldi Napoli, Napoli, Campania
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l - PPDS, Meldola, Forli-Cesena
  - Istituto Nazionale Dei Tumori, Milan, Lombardy
  - Instituto Europeo Di Oncologia, Milan, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Centro Di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Santa Maria Delle Croci, Ravenna
- Japan (12):
  - Fujita Health University Hospital, Toyoake-Shi, Aiti
  - National Cancer Center Hospital East, Kashiwa-Shi, Chiba
  - Ehime University Hospital, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Miyagi Cancer Center, Natori-shi, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka International Cancer Institute, Chuo Ku, Osaka
  - Saitama Cancer Center, Komoro, Saitama
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
- VU Medisch Centrum, Amsterdam, North Holland, Netherlands
- Portugal (5):
  - Centro Hospitalar do Porto Hospital de Santo Antonio, Santa Maria da Feira, Aveiro District
  - Hospital Cuf Porto, Vila Nova de Gaia, Porto District
  - Centro Hospitalar de Lisboa Norte E.P.E Hospital Pulido Valente, Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
  - Centro Hospitalar de Sao Joao, E.P.E., Porto
- Russia (2):
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg, Leningradskaya Oblast'
  - LLC "EuroCityClinic", Saint Petersburg, Sankt-Peterburg
- National Cancer Centre, Singapore, Singapore
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
- Spain (10):
  - ICO lHospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario A Coruna, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Karolinska Universitetssjukhuset Solna, Stockholm, Södermanland County, Sweden
- Taiwan (9):
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Dalin
  - National Taiwan University Hospital - YunLin Branch, Douliu
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Baskent University Medical Faculty Adana Practice and Research Center, Yüreğir, Adana
  - T.C. Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Kadıköy, Istanbul
  - Ege University Medical Faculty, Bornova, İzmir
  - SAKARYA University Medical Faculty, Karaman, Sakarya
  - Hacettepe University Medical Faculty, Ankara
  - Trakya University Medical Faculty, Edirne
- Ukraine (3):
  - Municipal Non-profit Enterprise "City Clinical Hospital # 4" of Dnipro City Council - PPDS, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv, Kharkivs’ka Oblast’
  - Private Enterprise Private Manufacturing Company Acinus, Kropyvnytskyi
- United Kingdom (5):
  - University College London Hospitals (UCLH), London, London, City of
  - Royal Marsden Hospital - Surrey, Sutton, Surrey
  - Clatterbridge Centre For Oncology, Bebington, Wirral
  - Leicester General Hospital, Leicester
  - The Christie NHS Foundation Trust - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Janne PA, Wang BC, Cho BC, Zhao J, Li J, Hochmair M, Peters S, Besse B, Pavlakis N, Neal JW, Kato T, Wu YL, Nguyen D, Lin J, Lin J, Vranceanu F, Szumski A, Lin HM, Fram RJ, Mok TSK. First-Line Mobocertinib Versus Platinum-Based Chemotherapy in Patients With EGFR Exon 20 Insertion-Positive Metastatic Non-Small Cell Lung Cancer in the Phase III EXCLAIM-2 Trial. J Clin Oncol. 2025 May;43(13):1553-1563. doi: 10.1200/JCO-24-01269. Epub 2025 Jan 29. PMID 39879577